CLINICAL TRIAL: NCT02329002
Title: Multicenter Implementation of MR Imaging Studies in Irradiated Hereditary Retinoblastoma Survivors for Assessment of the Value of Craniofacial MRI Screening for Early Detection of Second Craniofacial Primary Tumors and to Enhance Survival
Brief Title: SPT Screening in Irradiated Hereditary Retinoblastoma Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ODAS (Unknown)
Responsible Party: Principal Investigator, Marcus de Jong, Mr., Amsterdam UMC, location VUmc
Other Study IDs: Rb-SPT-SCR
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; Second primary tumor; Screening; Magnetic resonance imaging
MeSH Terms: conditions — Retinoblastoma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magnetic resonance imaging — MR imaging protocol should include a thin-slice (3-4 mm) short TI inversion recovery (STIR) sequence or fat-saturated T2-weighted images in axial direction. Furthermore, a 3D-T1 weighted sequence with isotropic voxels will be obtained, with reconstruction in 3 directions. If suspicious lesions are detected, additional MR imaging has to be performed, including contrast-enhanced images.

SUMMARY:
Rationale: Hereditary retinoblastoma survivors have an increased risk to develop second primary tumors (SPT) at a later age (with the highest risk in their teens), especially when they have been irradiated for retinoblastoma. The investigators hypothesize that regular screening with magnetic resonance imaging (MRI) could lead to early detection of SPTs leading to improved survival.

Objective: To evaluate the potential benefit of craniofacial MRI screening for early detection subclinical secondary cancers in patients previously irradiated for hereditary retinoblastoma.

Study design: Prospective multicenter non-invasive screening study. The total study duration will be four years of screening plus five years of follow-up.

Study population: Irradiated hereditary retinoblastoma patients 8-18 years old Main study parameters/endpoints: To evaluate the ability of craniofacial MRI for early detection of SPTs, the investigators will determine the sensitivity and specificity of MRI at detecting SPTs in irradiated hereditary retinoblastoma patients.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Included patients will undergo yearly craniofacial MRI for a period of 4 years. They will also be asked to fill out a psychological burden assessment form each visit. A potential risk of screening might be associated anticipatory anxiety, but screening also could be reassuring for patients and their parents; the investigators are not sure which will outweigh. False-positive results from MRI screening could lead to unnecessary further diagnostics leading to possible added anxiety and diagnostics (e.g., biopsies). However, this group of patients have a high risk of developing SPTs, with poor 5-year survival statistics. Early detection and therefore treatment of earlier stage (smaller) tumors, might therefore increase survival of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of hereditary retinoblastoma
* Patients that have been treated with external beam radiotherapy for retinoblastoma
* Age of patients at the first MR scan: 8 years or older (≥8 years old), but only as soon as the MR scan can be performed without sedation or general anesthesia, and until and including 18 years of age (≤18 years old).

Exclusion Criteria:

* MRI related exclusion criteria:

  * Claustrophobia
  * Foreign non MR compatible metal objects in the body
  * Foreign incompatible metal objects in or close to the head
  * Exclusion criterium for additional contrast sequences: Allergic reaction to contrast administration in the past

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The potential study population will be irradiated hereditary retinoblastoma survivors in the Netherlands and joining centers from other countries. Currently, there is no screening program for these high-risk patients. The age of patients at highest risk of developing craniofacial SPTs is 8-18 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of MRI for the detection of second primary tumors in hereditary irradiated retinoblastoma | 4 years
  The primary objective of the study is to evaluate the benefit of early detection of craniofacial second primary tumors with MRI in previously irradiated hereditary retinoblastoma survivors. The main outcome measure for assessing the benefit of screening will be the diagnostic accuracy of MRI for detecting craniofacial SPTs: sensitivity (true-positive and false-negative results) and specificity (true-negative and false-positive results).

SECONDARY OUTCOMES:
5-year survival | 9 years
  A secondary objective is to assess the 5-year survival of second primary tumors (SPT) found by screening, SPTs missed by screening, and the non-SPT patients
Descriptive statistics | 4 years
  Recording and monitoring location and characteristics (clinical, radiological, histological, treatment) of patients with SPTs: total number of patients included, median follow-up time + range, number of asymptomatic SPTs detected by screening, number of symptomatic SPTs missed by screening, number of SPTs developed after the end of screening, number of SPTs that were totally resected, location of tumor, type of tumor, size of tumor
Feasability assessment | 4 years
  Assessment of the feasibility of such this screening program: (a) percentage of patients (or family) willing to participate; (b) compliance of patients and their families to the screening program
Assessing the psychosocial burden or benefit | 4 years
  Once a year during the visits, the patient will be asked to fill out the Hospital Anxiety and Depression Scale (HADS).

CONTACTS AND LOCATIONS:
Overall Officials: Jonas A Castelijns, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands